CLINICAL TRIAL: NCT07026045
Title: Effects of Post Isometric Relaxation Versus Post Facilitation Stretch Techniques on Pain, Mobility and Disability in Patients With Chronic Low Back Pain
Brief Title: Post Isometric Relaxation Versus Post Facilitation Stretch Techniques in Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rao Irfan- REC/RCR&AHS 24/0136
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: Low back pain; Post isometric relaxation; Post facilitation stretch
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Post isometric relaxation (Lewit,s)
  Interventions: Other: Post isometric relaxation (Lewit,s)
- Group B (Active Comparator): Post facilitation stretch (Janda's technique)
  Interventions: Other: Post-Facilitation Stretch Technique (Janda's technique)

INTERVENTIONS:
Other: Post isometric relaxation (Lewit,s) — Post-isometric relaxation technique for the erector spinae, Iliopsoas, Quadratus Lumborum
  Arms: Group A
Other: Post-Facilitation Stretch Technique (Janda's technique) — Post-Facilitation Stretch Technique for the erector spinae, Iliopsoas, Quadratus Lumborum
  Arms: Group B

SUMMARY:
This randomized controlled trial will be conducted at Riphah Rehabilitation Clinic and Spinacure clinic in Lahore over a 9-month period. A sample size of 42 participants, aged 18 to 45, will be selected using convenient sampling. Informed consent will be obtained from all participants. Participants will be divided into two groups: Group A will receive Post-Isometric Relaxation in addition to standard physical therapy, while Group B will receive Post-Facilitation Stretch in addition to standard physical therapy. Outcome measures, including the Numeric Pain Rating Scale (NPRS) for pain, inclinometer for mobility assessment, and Oswestry Disability Index (ODI) Urdu version for disability, will be assessed at baseline and after 4 weeks. Inclusion criteria include patients with CLBP aged 18-45 years, with pain levels between >3 and <7 on the NPRS, and an ODI score between 14% and 50%. Exclusion criteria include any neurological symptoms, systemic soft tissue and bony disease, and previous spinal surgeries. Data will be analyzed using IBM SPSS 25.0.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the primary causes of physical impairment globally, affecting a significant portion of the population. It is associated with a high rate of absenteeism from work and substantial healthcare costs due to its pervasive nature. Chronic low back pain (CLBP), specifically, is a condition where pain is localized in the lumbar region and persists for more than 12 weeks. In contrast to acute low back pain, which typically resolves within six weeks, CLBP is characterized by a complex interplay of physical, psychological, and social factors that contribute to its persistence and chronicity .

Compared to other diseases, it is the primary cause of medical consultations, affects quality of life and performance at work, and occurs in a proportion that is similar in all cultures and ethnicities. Over 20% of people globally suffer from chronic LBP, and 24-80% of individuals experience a relapse during the first year. The prevalence of chronic low back pain (CLBP) in Pakistan is a significant health concern. A national survey conducted in 2021 found that 18% of individuals experiencing chronic pain reported low back pain as their primary complaint. This survey, involving 4,801 participants, highlighted the substantial impact of CLBP on daily life and the need for better pain management and awareness among patients (Journal of the Medical Association).

Management of CLBP typically involves a combination of pharmacological and non-pharmacological treatments. Pharmacological interventions include nonsteroidal anti-inflammatory drugs (NSAIDs), muscle relaxants, and analgesics to manage pain and inflammation. In some cases, antidepressants and anticonvulsants are prescribed for their pain-modulating effects. Non-pharmacological approaches are crucial for improving mobility and function. Physical therapy, including exercise programs designed to strengthen core muscles and improve flexibility, plays a vital role in rehabilitation. Manual therapy techniques, such as spinal manipulation and massage, and cognitive-behavioral therapy (CBT) to address the psychological aspects of chronic pain are also important. Lifestyle modifications, such as weight management, ergonomic adjustments, and activity modifications, are essential components of a comprehensive treatment plan.

Chronic low back pain (CLBP) is a prevalent and serious problem that affects millions of people, disrupting their daily activities and quality of life. To manage this condition effectively, strategies that reduce pain, improve movement, and lessen disability are needed. Post Isometric Relaxation (PIR) and Post Facilitation Stretch (PFS) are two techniques that can help with these goals. This study aims to compare the effects of PIR and PFS on pain, mobility, and disability in patients with CLBP. By finding out which method is more effective, clinicians can choose better treatments, improve patient outcomes, create better treatment guidelines, and enhance the quality of life for those suffering from chronic low back pain. This approach can also help lower healthcare costs by reducing the need for more invasive treatments and long-term medication use.

ELIGIBILITY:
Inclusion Criteria:

* Age of patient between 18 to 45 year
* Both gender
* (LBP) for more than 3 months
* Diagnosis of Chronic Low Back Pain (CLBP)
* Negative SLR, negative faber test, negative lumber quadrant
* Lumber extension test positive, positive scobber test
* Having low back pain below the costal margin and above inferior gluteal folds and suffering from low back pain
* Disability level of more than 14% and less than 50% according to Oswestry questionnaire
* NPRS score of >3 to ≤7

Exclusion Criteria:

* Chronic systemic soft tissue and bony disease
* Any neurological symptoms involving Prolapsed Intervertebral Disc, Radiculopathy Back pain with trauma
* History of recent abdominal, back surgeries and pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Baseline, 4th Week
Lumbar Flexion | Baseline, 4th Week
Lumbar Extension | Baseline, 4th week
Lumbar Side Flexion | Baseline, 4th Week
Oswestry Disability Index | Baseline, 4th Week

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Tulder MW, Koes BW, Bouter LM. Conservative treatment of acute and chronic nonspecific low back pain. A systematic review of randomized controlled trials of the most common interventions. Spine (Phila Pa 1976). 1997 Sep 15;22(18):2128-56. doi: 10.1097/00007632-199709150-00012. PMID 9322325
- [Background] Amjad MA, Siddiqui AM, Bashir K, Ghafoor AU, Durrani RS. Prevalence of chronic pain in Pakistan - a national survey. J Pak Med Assoc. 2023 Jun;73(6):1217-1220. doi: 10.47391/JPMA.6671. PMID 37427618
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886